CLINICAL TRIAL: NCT03532048
Title: Adapting and Assessing the Feasibility Of 'Healthy Dads Healthy Kids' For US Latinos
Brief Title: Feasibility of Healthy Dads Healthy Kids Latino
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Teresia O'Connor, Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-38237; R34HL131726 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-05-22 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Feasibility
Keywords: Hispanic; Fathers; Child; Obesity Prevention; Cultural adaptation; Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Feasibility study with a randomized wait-list control group design
Masking Description: In this feasibility study there will be no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Papás Saludables, Niños Saludables Program
  Interventions: Behavioral: The Papás Saludables, Niños Saludables Program
- Wait-list Control (Other): The Papás Saludables, Niños Saludables Wait-list Control
  Interventions: Behavioral: The Papás Saludables, Niños Saludables Wait-list Control

INTERVENTIONS:
Behavioral: The Papás Saludables, Niños Saludables Program — Papás Saludables, Niños Saludables is a 10 week program for fathers and their children that meets weekly. Each session is 90 minutes long: 15 min introduction, 30 min pull-out sessions for fathers and children, and 45 min active play sessions together. Fathers are encouraged to improve their eating and physical behaviors to lose weight and to be healthy role models for their child. Children are encouraged to help their fathers lose weight and improve their health. The program has been adapted to contextualize the information for low-income Hispanic families and changed to US food and physical activity guidelines. Mothers will be provided a Handbook and will be sent short videos, recipe links, and short motivational messages every week covering the same topics as in the sessions.
  Other Names: Culturally adapted Healthy Dads Healthy Kids Program
  Arms: Intervention Group
Behavioral: The Papás Saludables, Niños Saludables Wait-list Control — The same program as above delivered to the wait-list control after the T1 follow-up data has been collected.
  Arms: Wait-list Control

SUMMARY:
This is a feasibility study of a culturally adapted version of Healthy Dads Healthy Kids for Hispanic families. The adapted version called Papás Saludables, Niños Saludables is a father-targeted program for child obesity prevention and weight loss for fathers. The feasibility study will be conducted with 40 Hispanic families. Baseline assessments (T0) will be completed on all participating family members, followed by randomization to start the program immediately (intervention group), or 6-7 months later (wait-list control). Post assessments (T1) will be completed on the full sample once the intervention group has participated in the 10 week Papás Saludables, Niños Saludables program. A process evaluation will be conducted to assess the feasibility outcomes of the study.

DETAILED DESCRIPTION:
This is a feasibility study of a culturally adapted version of Healthy Dads Healthy Kids for Hispanic families, called Papás Saludables, Niños Saludables. It is a father-targeted program for child obesity prevention and weight loss for fathers. The feasibility study will be conducted with 40 Hispanic families at a large community pediatric clinic serving children with Medicaid or CHIP. Enrollment will include fathers, their 5-11 year old child(ren) and their co-parent (e.g. mother) as a family unit (anticipate 160 individuals). Fathers and their child(ren) will be the primary target in the study, but mothers also participate, if available. Multiple children per family can enroll if they meet the inclusion/exclusion criteria, but families will be encouraged to limit the number of children who participate to no more than three. Fathers will be screened for their health to participate in the physical activity portion of the study and whether they meet inclusion/exclusion criteria. The health screening will follow the 2015 updated American College of Sport Medicine exercise pre-participation screening protocol. Fathers who otherwise qualify, but do not pass the health screener will be provided a letter to be seen by their PCP to obtain clearance for exercise participation. If they do not have a PCP they will be instructed to contact their health insurance for a list of doctors and if they do not have health insurance, a list of sliding scale clinics will be provided.

Once screened, consented and enrolled, baseline data will be collected on the fathers, children and mothers. Data assessments include demographics, height, weight, and waist circumference on fathers and children, blood pressure and heart rate on fathers, physical activity and sleep on fathers and children (as measured by wearing accelerometers for 5-7 days), screen media use by survey questions of fathers and children, dietary intake on fathers and children (by food frequency questionnaires), food and physical activity parenting practices, co-parenting alliance scale, acculturation (Bi-Acculturation Scale), respeto (Respect sub-scale from the Mexican-American Cultural Values scale) and Pan-American familism scale on fathers and mothers. Mothers, if available, will be asked to assist the child in completing their questionnaires. If the family consists of a single father, he will assist the child in completing their questionnaires. Fathers and children will be instructed in wearing their accelerometer and told to wear it 24 hours/day for the next 7 days, only taking it off when there is potential for getting it wet (e.g. bathing, showering, swimming). Study staff will remind the father and child to wear their monitor by text, email or phone call (depending on family preference) several times during week. Accelerometers and wear logs can be returned at the clinic or by prepaid envelope provided by the study. Once received back, accelerometer data will be reviewed for completeness (minimum of 8 hours/day for 5 days including 2 weekend days). If accelerometer data is not complete, the father and/or child will be given the option to wear the monitor for additional days to complete the data.

After baseline data are collected, families will be stratified into preferred language of program (English or Spanish) and randomly assigned to receive the program immediately (Intervention Group, N=20) or after a 5-7 month wait list period (Wait-list Control group, N=20).

After the 10 session program is completed, post-assessment data will be collected on all 40 families in the same way as described for the baseline data collection. In addition, fathers, mothers and children who took part in the Papás Saludables, Niños Saludables program will be asked to complete a satisfaction survey. Families who were assigned to the control group will start the program after the second data collection. Data collection on the wait-list control group will only consist of weight, height, and satisfaction survey.

Exit interviews of a sub-sample of fathers, mothers and children each who took part in the Papás Saludables, Niños Saludables program will be conducted. The interviews will be audio-recorded and coded for themes.

Process Evaluation: Recruitment, screening and enrollment will be tracked by study staff. Attendance to the data collection sessions and HDHK program sessions will be tracked by the program facilitators and research staff. Fidelity of program delivery by the facilitator will be assessed via research staff observation and use of a delivery checklist for each session.

ELIGIBILITY:
Inclusion Criteria:

* Latino/Hispanic fathers, mothers (if available) over the age of 18, with at least one healthy child between the ages 5-11 years old, and target child between the ages of 5-11 years old
* Child is a patient at one of the TCHP Center for Children and Women Clinics
* Parents able to read and write in either Spanish or English
* Latino/Hispanic families who live in the Greater Houston area
* Fathers and children willing to wear an accelerometer for a 7 day study period at baseline and 4 months later
* Fathers with a BMI > 25 and <40
* Fathers pass the American College of Sports Medicine (ACSM) health screener to participate or get medical clearance to participate from a medical doctor.

"Father" will be defined as an adult "father figure" in the child's life. This can include a biological father, step father, adapted father, grandfather, older adult brother, uncle or other male figure who is a father figure for the child and helps with caring/raising the child.

Exclusion Criteria:

* Child or parent with a disease affecting their dietary intake (severe GI disease or multiple food allergies), physical activity behaviors (e.g., physical disability, severe asthma), cognitive functioning (e.g., Down's syndromes, Fragile X), or psychiatric functioning (e.g. schizophrenia in parent)
* Plans of moving away from Harris County in the next year
* Fathers BMI>40
* Fathers who have lost more than 10 pounds recently, are in a current weight loss program or taking medications to lose weight
* Fathers who fail ACSM health screening and do not provide a MD letter approving participation in the program.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Latino/Hispanic fathers over the age of 18, with at least one healthy child between the ages 5-11 years old, and a target child between the ages of 5-11 years old who attends the TCHP Center for Children and Women Clinics in Houston, TX are eligible
Enrollment: 160 (Actual)
Dates: Start 2018-08-11 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresia O'Connor, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- TCHP The Center for Children and Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan PJ, Lubans DR, Callister R, Okely AD, Burrows TL, Fletcher R, Collins CE. The 'Healthy Dads, Healthy Kids' randomized controlled trial: efficacy of a healthy lifestyle program for overweight fathers and their children. Int J Obes (Lond). 2011 Mar;35(3):436-47. doi: 10.1038/ijo.2010.151. Epub 2010 Aug 10. PMID 20697417
- [Background] Morgan PJ, Collins CE, Plotnikoff RC, Callister R, Burrows T, Fletcher R, Okely AD, Young MD, Miller A, Lloyd AB, Cook AT, Cruickshank J, Saunders KL, Lubans DR. The 'Healthy Dads, Healthy Kids' community randomized controlled trial: a community-based healthy lifestyle program for fathers and their children. Prev Med. 2014 Apr;61:90-9. doi: 10.1016/j.ypmed.2013.12.019. Epub 2013 Dec 29. PMID 24380796
- [Background] Riebe D, Franklin BA, Thompson PD, Garber CE, Whitfield GP, Magal M, Pescatello LS. Updating ACSM's Recommendations for Exercise Preparticipation Health Screening. Med Sci Sports Exerc. 2015 Nov;47(11):2473-9. doi: 10.1249/MSS.0000000000000664. PMID 26473759
- [Background] O'Connor TM, Beltran A, Musaad S, Perez O, Flores A, Galdamez-Calderon E, Isbell T, Arredondo EM, Parra Cardona R, Cabrera N, Marton SA, Baranowski T, Morgan PJ. Feasibility of Targeting Hispanic Fathers and Children in an Obesity Intervention: Papas Saludables Ninos Saludables. Child Obes. 2020 Sep;16(6):379-392. doi: 10.1089/chi.2020.0006. Epub 2020 May 28. PMID 32466678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Goal of 40 families (160 individuals) to be recruited.
Units Other Than Participants: families
Period: Overall Study
Arm/Group | Intervention Group | Wait-list Control
Started | 68; 19 families (68 individuals (19 fathers, 31 children & 18 mothers)) | 67; 17 families (67 individuals (17 fathers, 33 children & 17 mothers))
Completed | 49; 14 families (49 individuals (14 fathers, 22 children, 13 mothers). 1 father only took part in interview) | 50; 13 families (50 individuals (13 fathers, 24 children & 13 mothers))
Not Completed | 19; 5 families | 17; 4 families
Not completed — Lost to Follow-up | 12 | 17
Not completed — Withdrawal by Subject | 7 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: families
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Wait-list Control | Total
Number analyzed (Participants) | 68 | 67 | 135
Number analyzed (families) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was not collected on mothers. Population: Age reported separately for fathers and children. Age was not collected on the mothers.
  years
    Fathers: number analyzed (Participants) | 19 | 17 | 36
    Fathers | 36.8 (7.61) | 36.1 (5.25) | 36.5 (6.52)
    Children: number analyzed (Participants) | 31 | 33 | 64
    Children | 8.8 (2.26) | 8.1 (1.96) | 8.5 (2.12)
    Mothers: number analyzed (Participants) | 18 | 17 | 35
    Mothers | NA (NA) — age not collected for mothers | NA (NA) — age not collected for mothers | NA (NA) — age not collected for mothers
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 37 | 71
  Male | 34 | 30 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic : Fathers | 19 | 17 | 36
  Hispanic : Children | NA — Not asked | NA — Not asked | NA — Total not calculated because data are not available (NA) in one or more arms.
  Hispanic : Mothers | NA — Not asked | NA — Not Asked | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Retention of Subjects in Study Assessments
Description: Retain 80% of intervention and control participants for pre- and post-assessments
Time Frame: 5 months
Population: families
Measure: Number; unit: families
Units Other Than Participants: families
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 68 | 67
Number analyzed (families) | 19 | 17
families | 14 | 13

2. Primary Outcome: Recruitment of Subjects Into Study
Description: Recruitment criteria was to recruit 40 Latino fathers and their families in ≤ 4 months. The actual recruited number of fathers with their family is reported as the outcome withe the percentage of goal achieved (actual/goal).
Time Frame: 4 months
Population: The goal was to recruit 40 families (20 for intervention group and 20 for wait-list control group) in </=4 months.
Measure: Count of Units; unit: families
Units Other Than Participants: families
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 20 | 20
Number analyzed (families) | 20 | 20
families | 19 | 17

3. Primary Outcome: Subject Attendance to Program Sessions
Description: Attendance of families to the 10 PSNS program sessions were recorded each week for the intervention group and later the wait-list control group. The goals was to maintain ≥70% attendance to program sessions
Time Frame: 10 weeks
Population: Families were the unit of analysis
Measure: Mean (Standard Deviation); unit: sessions attended
Units Other Than Participants: families
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 19 | 17
Number analyzed (families) | 19 | 17
sessions attended | 5.6 (4.1) | 5.6 (3.8)

4. Secondary Outcome: Percentage of Fathers and Mothers Who Reported Their Satisfaction With the PSNS Program as Excellent to Good on the "Healthy Dads Healthy Kids Satisfaction Survey"
Description: The participating Latino fathers will be satisfied with the program as measured by 80% 'excellent'-'good' satisfaction from questionnaires and exit interviews with the Latino fathers and their co-parent (typically children's mother).
Time Frame: 10 weeks
Population: parent (fathers and mothers) who reported "excellent" or "good" on 5-point scale.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 24 | 23
Participants | 24 | 23

5. Secondary Outcome: Data Collection Completeness
Description: Ability to collect anthropometric, behavioral and parenting data on at least 75% of the Latino fathers and anthropometric, and behavioral data on their children (both groups) at baseline and follow up
Time Frame: 5 months
Population: families
Measure: Count of Units; unit: families
Units Other Than Participants: families
Arm/Group | Intervention Group | Wait-list Control
Number analyzed (Participants) | 68 | 67
Number analyzed (families) | 19 | 17
families | 13 | 13

ADVERSE EVENTS:
Time Frame: 3 months during the intervention
Description: Reviewed by staff weekly during intervention delivery. Definitions same as in clinicaltrial.gov
  Clarification:
  minor injury (superficial scrape), time-limited tiredness, fatigue, or dry mouth immediately after exercise portion of intervention not considered adverse event, but anticipated with exercise.
Arm/Group | Intervention Group | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67
Other Adverse Events (participants affected / at risk) | 0/68 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT03532048/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT03532048/ICF_001.pdf